CLINICAL TRIAL: NCT06720441
Title: Predictors of Improvement and Deterioration of Community Acquired Pneumonia in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Nageh Thabet Eshak, MNTEshak, Assiut University
Other Study IDs: Pneumonia prognosis in child
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-09

CONDITIONS: Predictors of Improvement and Deterioration of Community Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Predictors of improvement and deterioration of community acquired pneumonia in children Community-acquired pneumonia (CAP) is the most prevalent respiratory infectious disease. It is defined as an acute infection of the lung parenchyma that is acquired outside the hospital. Community-acquired pneumonia (CAP) is one of the most common disorders faced in clinical practice . [1,2] Childhood CAP is the leading cause of death in children younger than five years globally[3] .

Acute phase reactants (APR) are inflammatory mediators that show significant alternations in serum levels in response to inflammation, these markers are responsible for some adverse effects such as anorexia, fever, fatigue, and anemia of chronic illness [4] APR can be applied for the assessment of disease severity in CAP in collaboration with clinical evaluation and pneumonia severity scores [5]. The most common APR are (NLR), CRP, and ESR, changes in the level of these indices can be used in the diagnosis and prognosis of inflammatory and infectious diseases [5] NLR is a rapid, simple, and cheap maker of the systemic inflammatory process, it is calculated as the ratio between neutrophil count to lymphocyte count from peripheral blood sample. Numerous researches have assessed the role of NLR in many infectious diseases such as sepsis, bacteremia, and septic shock, in addition, it can predict the severity and outcome of CAP [6] CRP is one of the best indicators of the acute phase response to inflammation. This serum protein is synthesized by hepatocytes and is classified as an acute-phase protein based on its increased serum concentration during inflammation and infection[7] So, the aim of the current study was to assess levels of APR such as total leucocytic count (TLC), platelets, neutrophils, neutrophils-to-lymphocyte ratio (NLR), CRP, D-dimer, Ferritin, and ESR in patients with CAP (as a primary outcome) and to correlate between their measured values and disease severity (as a secondary outcome)

DETAILED DESCRIPTION:
Assessment of community-acquired pneumonia (CAP) severity in association with various pneumonia severity scores. So, the aim of the study was to assess levels of APR such as total leucocytic count (TLC), platelets, neutrophils, neutrophils-to-lymphocyte ratio (NLR), CRP, D-dimer, ferritin, and ESR in patients with CAP and to correlate between their values and disease severity.

ELIGIBILITY:
Inclusion Criteria All patients above a month and below 18 years old, both sexes, fulfilling diagnosis of CAP

Exclusion Criteria:

* Non-pulmonary infections, liver, renal, and cardiac diseases.and neonates with age less than a month

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inclusion Criteria All patients above a month and below 18 years old, both sexes, fulfilling diagnosis of CAP
  Exclusion Criteria:
  * Non-pulmonary infections, liver, renal, and cardiac diseases.and neonates with age less than a month
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Relation between acute phase reactants and pneumonia | 1 year
  Assess levels of APR such as total leucocytic count (TLC), platelets, neutrophils, neutrophils-to-lymphocyte ratio (NLR), CRP, D-dimer, Ferritin, and ESR in patients with CAP (as a primary outcome)

SECONDARY OUTCOMES:
Predictors of improvement and deterioration of community acquired pneumonia in children | 1 year
  Predictors of improvement and deterioration of community acquired pneumonia in children

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: 1. — https://ejb.springeropen.com/articles/10.1186/s43168-023-00234-1